CLINICAL TRIAL: NCT06538753
Title: Silver Leaf During Pregnancy in French Guiana : Use and Impact on Health
Acronym: Feydarjan
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: Fey darjan
Record Dates: First submitted 2024-07-18; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy Complications; Herbal Medicine Adverse Reaction
Keywords: Pregnancy; Traditional medecine use; Traditional medecine adverse reaction; Silver leaf; French Guiana
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive, observational, cross-sectional study among women who have given birth in one of French Guiana's maternity hospitals to determine if the use of silver leaf is frequent and could have an impact on pregancy outcomes. This Fey darjan project is an ancillary study of the Nutri Pou Ti'Moun 1 project

DETAILED DESCRIPTION:
French Guiana's ethnomedicines use is still very dynamic, with a significant level of herbal medicine use per inhabitant (17.6 citations of use per inhabitant surveyed) and the continual integration of new species into the local medicinal flora. Over a period of 30 years, studies noted significant changes and mutations in plant-based care methods, favored by a significant intercultural mix (close border areas and migrant population from the Caribbean and South America).

The species Ocotea guianensis Aublet (Lauraceae), known in French Guiana as 'feuille d'argent' (féy darjan in Creole, silvon leaf in english), is used locally to facilitate childbirth. This use (a decoction of leaves administered to parturients as a sitz bath) among the Palikur (an indigenous Amerindian people from northern Amapá in Brazil and eastern French Guiana) and coastal Creoles. This use has been observed more recently by Tareau (2020) among Haitian and Guyanese Creole women According to a preliminary study by a perinatal network in French Guiana, cases of acute foetal distress at the time of delivery and post-partum haemorrhage have been observed in pregnant women who have used silver leaf decoctions, without a statistical or pathophysiological link being formally established.

From an epidemiological point of view, the frequency of use of Silver Leaf Decoctions (SLD) and the medical consequences of this use during childbirth and the immediate post-partum period have not been quantified in French Guiana. Although health-care providers have observed that some women use SLDs when certain pathological events occur during childbirth, no study has demonstrated a definite link between SLDs and complicated childbirth.

The profile of users, the ways in which SLDs are used during pregnancy, and their impact on childbirth, uterine contractions and the immediate post-partum period also need to be clarified. The perception and representations of this practice from the point of view of caregivers are also elements to be taken into consideration.

The research hypothesis is that the use of silver leaf by parturients in French Guiana is frequent and could have an impact on pregnancy outcomes (prolonged labor, ineffective contractions, perinatal pain, cardio-fetal rhythm abnormalities, post-partum hemorrhage...).

ELIGIBILITY:
Inclusion Criteria:

* Women admitted for delivery in one of the French Guiana maternity hospitals and previsouly included in the study Nutri Pou Ti Moun 1 (NCT05653128)

Exclusion Criteria:

* Refusal to participate to study or absence of collection of non-opposition of participant
* Lack of parental consent for minor participants
* Women under gardianship or curatorship

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women delivering in one of the French Guiana maternity hospitals and previously included in study Nutri Pou Ti Moun 1
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of silver leaf decoction use | At inclusion
  To estimate the prevalence of silver leaf decoction use among women who gave birth in one of the French Guiana maternity hospitals assessed by a questionnaire

SECONDARY OUTCOMES:
Description of pregnancy outcomes | At inclusion
  To describe pregnancy outcomes of women using SLDs in the prenatal period in relation to perinatal indicators in French Guiana (gestational diabetis, hypertension, pre-eclampsia/eclampsia, foetal weight abnormalities ), documented from medical file
Description of immediate post-partum outcomes | At inclusion
  To describe immediate post-partum outcomes of women using SLDs in the prenatal period in relation to perinatal indicators in French Guiana (vaginal delivery, C-section, post-partum bleeding, foetal cardio rhythm abnormalities...), documented from medical file
Description of delivery pain management method | At inclusion
  To describe the delivery pain management method of women using SLDs in prenatal period in relation to women not using SLDs (no delivery pain management method, epidural, spinal analgesia, general anaesthetic) documented from medical file
Use and representations of women using SLDs | At inclusion
  To describe how women use SLDs during delivery assessed by a questionnaire
Health professionals comprehensions on SLDs use during delivery | At inclusion
  To describe the comprehensions of health professionals on SLDs use during delivery assessed by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Celia BASURKO, MD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang CW, Ko FN, Su MJ, Wu YC, Teng CM. Pharmacological evaluation of ocoteine, isolated from Cassytha filiformis, as an alpha 1-adrenoceptor antagonist in rat thoracic aorta. Jpn J Pharmacol. 1997 Mar;73(3):207-14. doi: 10.1254/jjp.73.207. PMID 9127815
- [Background] Antonio ADS, Aguiar ATC, Dos Santos GRC, Pereira HMG, da Veiga-Junior VF, Wiedemann LSM. Phytochemistry by design: a case study of the chemical composition of Ocotea guianensis optimized extracts focused on untargeted metabolomics analysis. RSC Adv. 2020 Jan 21;10(6):3459-3471. doi: 10.1039/c9ra10436d. eCollection 2020 Jan 16. PMID 35497754
- [Background] Antonio AS, Veiga-Junior VF, Wiedemann LSM. Ocotea complex: A metabolomic analysis of a Lauraceae genus. Phytochemistry. 2020 May;173:112314. doi: 10.1016/j.phytochem.2020.112314. Epub 2020 Feb 29. PMID 32120118
- [Background] Guterres Zda R, da Silva AF, Garcez WS, Garcez FR, Fernandes CA, Garcez FR. Mutagenicity and recombinagenicity of Ocotea acutifolia (Lauraceae) aporphinoid alkaloids. Mutat Res. 2013 Sep 18;757(1):91-6. doi: 10.1016/j.mrgentox.2013.07.004. Epub 2013 Jul 24. PMID 23892138
- See also: Traditional pharmacopoeia in Frecnh Guiana — http://www.editions.ird.fr/produit/278/9782709923453/pharmacopees-traditionnelles-en-guyane
- See also: Plants of love : ethnobotany of plant species used for sexual purposes in Afro-descendant communities in French Guiana — http://www.ethnopharmacologia.org/boutique/les-plantes-de-lamour-ethnobotanique-des-especes-vegetales-utilisees-autour-de-la-sexualite-dans-les-communautes-afro-descendantes-de-guyane-francaise-n63-20/
- See also: The hybrid pharmacopoeias of French Guiana : ethnobotany of a phytotherapy on the move — https://theses.hal.science/tel-02926473v1/file/These_Tareau_Marc_Alexandre.pdf